CLINICAL TRIAL: NCT06463964
Title: Predictors of Acute Kidney Injury in Patients With Acute Decompensated Heart Failure in Emergency
Status: Enrolling by invitation | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shady Medhat Farouk, Resident- Department of Internal Medicine, Sohag University
Other Study IDs: Soh-Med-24-05-17MS
Record Dates: First submitted 2024-06-04; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Acute Kidney Injury; Acute Heart Failure
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group I: ( Patients with worsening ADHF)
  Interventions: Diagnostic Test: Serum Creatinine
- Group II: (Patients with new (de novo ) ADHF)
  Interventions: Diagnostic Test: Serum Creatinine

INTERVENTIONS:
Diagnostic Test: Serum Creatinine — Laborataries for prediction of AKi in patients with ADHF
  Other Names: CBC; Estimated GFR; Lipid profile; Serum electrolytes; CKMB; Cardiac Troponin

SUMMARY:
Acute Decompensated Heart Failure ADHF is one of the leading causes of hospitalization. ADHF is a growing global health problem affecting more than 26 million individuals worldwide Acute Kidney Injury AKI is a common event in the natural disease history of patients with Heart Failure HF, The clinical importance of the co-existence of acute cardiac and renal dysfunction, known as acute cardiorenal syndrome CRS, and its management have recieved great attention recently Various studies have employed different criteria to define and calssify AKI. According to Risk, Injury, and Failure; and Loss, and End-stage kidney disease RIFLE criteria formulated by the Acute Dialyisis Quality Initiative ADQI AKI can be divided into five stages; renal injury risk, renal impairment, renal failure, renal function loss, and end stage kidney disease

DETAILED DESCRIPTION:
In the past few years, investigators have reported that AHF patients might experience "congestion", named to describe signs and symptoms of extracellular fluid accumulation that results in increased cardiac filling pressure. This triggers compensatory mechanisms such as the renin-angiotensin-aldosterone system, sympathetic nervous system, and other local mediators. These compensatory mechanisms interact to maintain fluid volume and "renal congestion" has been recognized as part of systemic congestion. Renal congestion, resulting from lower cardiac output, tubule glomerular feedback, increased intra-abdominal pressure and increased venous pressure, has been viewed as a contributor to renal function impairment in ADHF.

Most patients with acute CRS are treated in the emergency department ED. The findings provide important insight into the present situation of patients with ADHF who develop AKI in an emergency setting.

The current diagnostic paradigm for AKI relies largely on biomarkers of renal function (serum creatinine and urine output) that have been in clinical use for over 50 years but are known to be insensitive and slow to change after kidney injury . It is very important to detect kidney damage in the preclinical process with new diagnostic methods and thus to provide early intervention in AKI.

Changing AKI definition and classification by year, these existing prediction models also vary by population, region, sample size and research methods. However, many studies have found a high incidence of AKI and a large impact on outcomes in ADHF patients, data pooled from these studies are inadequate. So, we will conduct this study to evaluate predictors of AKI in patients with ADHF in emergency departments.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 Yrs Both Sexes Patients with ADHF

Exclusion Criteria:

* Patients udnergoing maintenance renal replacment therapy (RRT) such as hemodialysis and peritoneal dialysis History of CKD Kdiney transplantation Undergoing opeartions within 1 week before and after AKI events Drug Toxicity Rheumatologic or auto immune disease Acute infection Diretic therapy of radio-opaque contrast media in the last 15 days History of aminoglycosides, metformin and nonsteroid anti inflammatory drugs in the last 7 days Thyroid dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Aged >18 Yrs Both Sexes Patients with ADHF
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in serum creatinine in mg/dL in patients with acute decompensated heart failure in ER | 6 months
  Change in serum creatinine in patients with acute decompensated heart failure in ER

CONTACTS AND LOCATIONS:
Overall Officials: Magdy M Amin, Professor, Principal Investigator — Sohag University
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Afsar B, Ortiz A, Covic A, Solak Y, Goldsmith D, Kanbay M. Focus on renal congestion in heart failure. Clin Kidney J. 2016 Feb;9(1):39-47. doi: 10.1093/ckj/sfv124. Epub 2015 Nov 29. PMID 26798459
- [Background] Chahal RS, Chukwu CA, Kalra PR, Kalra PA. Heart failure and acute renal dysfunction in the cardiorenal syndrome. Clin Med (Lond). 2020 Mar;20(2):146-150. doi: 10.7861/clinmed.2019-0422. PMID 32188648
- [Background] Chen JJ, Lee TH, Kuo G, Yen CL, Chen SW, Chu PH, Fan PC, Chien-Chia Wu V, Chang CH. Acute Kidney Disease After Acute Decompensated Heart Failure. Kidney Int Rep. 2022 Jan 3;7(3):526-536. doi: 10.1016/j.ekir.2021.12.033. eCollection 2022 Mar. PMID 35257065
- [Background] Fuhrman DY, Stanski NL, Krawczeski CD, Greenberg JH, Arikan AAA, Basu RK, Goldstein SL, Gist KM; ADQI 26 workgroup. A proposed framework for advancing acute kidney injury risk stratification and diagnosis in children: a report from the 26th Acute Disease Quality Initiative (ADQI) conference. Pediatr Nephrol. 2024 Mar;39(3):929-939. doi: 10.1007/s00467-023-06133-3. Epub 2023 Sep 5. PMID 37670082